CLINICAL TRIAL: NCT01213069
Title: Staff Opinions and Knowledge Concerning Organ and Tissue Harvesting: an Investigation Among the Patient Care Personnel in the South-Mediterranean Region of France
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-I/2009/CB-01; 1391089 (Other: France: Commission Nationale de l'Informatique et des Libertés)
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Tissue and Organ Procurement
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all 5000 subjects: this is a purely descriptive study with one group
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The subjects are asked to fill out a questionnaire on the personal and professional situations, organ donation legislation, what happens in everyday practice, their own experience with donating their own organs, and what position they take.

SUMMARY:
The goal of this study is to evaluate the knowledge of paramedical and medical care personnel concerning organ and tissue donations, as well as their opinions on this activity.

ELIGIBILITY:
Inclusion Criteria:

* paramedical or medical care personnel from a participating center
* participates in organ donor activities
* works in a department with organ donor activity

Exclusion Criteria:

* personnel with no contact with organ donor activities
* personnel from non-participating centers
* refuses to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health care personnel in South-Mediterranean France
Sampling Method: Non-Probability Sample
Enrollment: 1859 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
VAS Negative/positive feeling | 1 day
  Visual Analog Scale from 0 to 100 where 0 is negative and 100 is positive.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Boutin, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (4):
- France (4):
  - AP-HM Hôpital Nord, Marseille
  - Hôpital Guy de Chauliac, CHU de Montpellier, Montpellier
  - Hôpital Cimiez, CHU de Nice, Nice
  - Centre Hospitalier Universitaire de Nîmes, Nîmes